CLINICAL TRIAL: NCT05248971
Title: Implementation of Trauma-focused Cognitive Behavioral Therapy (TF-CBT) in Norwegian Child and Adolescent Mental Health Clinics
Brief Title: Implementation of Truma-Focused Cognitive Behavioral Therapy (TF-CBT) in Norway
Acronym: TF-CBT
Status: Completed | Type: Observational
Sponsor: Norwegian Center for Violence and Traumatic Stress Studies (Other)
Responsible Party: Principal Investigator, Ane-Marthe Solheim Skar, PhD, Norwegian Center for Violence and Traumatic Stress Studies
Other Study IDs: TF-CBT 2012-2021
Record Dates: First submitted 2022-02-09; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: PTSD
Keywords: PTSD; Trauma treatment; Implementation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children screened for trauma and/or posttraumatic stress: Children were screened for trauma exposure and posttraumatic stress at one of the first meetings at the child and adolescent mental health clinic. For participants receiving TF-CBT, posttraumatic stress was also assessed during and after therapy.
  Interventions: Other: Trauma-focused cognitive behavioral therapy (TF-CBT)

INTERVENTIONS:
Other: Trauma-focused cognitive behavioral therapy (TF-CBT) — TF-CBT is an evidence-based treatment method for children and adolescents who have been exposed to trauma and experience posttraumatic stress symptoms. The treatment model has a family and caregiver focus, and non-offending caregivers are included in the treatment. TF-CBT is normally provided through 8-12 treatment sessions.

SUMMARY:
Trauma-focused cognitive behavioral therapy (TF-CBT) is an evidence-based treatment method for children and adolescents who have been exposed to traumatic experiences and who are experiencing posttraumatic stress symptoms. TF-CBT has been implemented in Norwegian child and adolescent mental health clinics since 2012. The Ministry of Health is funding the implementation project, and the Norwegian Center for Violence and Traumatic Stress Studies (NKVTS) is responsible for the implementation, including training of therapists, quality monitoring, and research.

DETAILED DESCRIPTION:
All participating child and adolescent mental health clinics received training by TF-CBT senior trainers at NKVTS in screening for trauma exposure and posttraumatic stress. A sub-sample of the therapists received training in TF-CBT. Data are collected on treatment outcomes for quality assurance.

ELIGIBILITY:
Inclusion Criteria:

* 6-18 years
* Referred to Norwegian child and adolescent mental health clinics

Exclusion Criteria:

* Below 6 years and above 18 years

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents aged 6-18 referred to Norwegian child and adolescent mental health clinics.
Sampling Method: Non-Probability Sample
Enrollment: 26500 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Child and Adolescent Trauma Screen (CATS) | 2012-2014
  Consists of two parts. Part 1 is a screening for exposure to potential traumatizing events; Part 2 is a screening for posstraumatic stress symptoms
Child PTSD Symptom Scale (CPSS) | 2015-2021
  Consists of two parts. Part 1 is a screening for exposure to potential traumatizing events; Part 2 is a screening for posstraumatic stress symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ane-Marthe S Skar, PhD, Principal Investigator — Norwegian Center for Violence and Traumatic Stress Studies

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Skar AS, Braathu N, Jensen TK, Ormhaug SM. Predictors of nonresponse and drop-out among children and adolescents receiving TF-CBT: investigation of client-, therapist-, and implementation factors. BMC Health Serv Res. 2022 Sep 29;22(1):1212. doi: 10.1186/s12913-022-08497-y. PMID 36175864